CLINICAL TRIAL: NCT06734299
Title: A Single-Center, Randomized, Clinical Study to Evaluate Usage of Facial Mineral Sunscreens With Differentiated Whitening Attributes in Multi-Cultural Skin Tones Through Instrumentation Measurements, Imaging, and Self-Assessments
Brief Title: A Study to Evaluate Usage of Mineral Sunscreens With Differentiated Whitening Attributes in Multi-Cultural Skin Tones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CS2024SK100197
Record Dates: First submitted 2024-12-12; First posted 2024-12-16 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-11

CONDITIONS: Sunscreen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sunscreen A (Experimental): At each visit, each enrolled subject will be randomly assigned 1 of the 3 Sunscreens to apply to both lower legs (between the knee and ankle) and then her full face. The subject will cleanse her hands with soap and water between the lower legs and face Sunscreen applications.
  After lower legs and facial Sunscreen applications are completed, a trained designee will delineate six 4 cm x 4 cm test sites on the subject's volar forearms (3 test sites per volar forearm). Then a trained designee will apply the assigned Sunscreen to the designated test sites in a consistent manner at a randomly assigned dose density of 0.25, 0.50, 0.75, 1.00, 1.50, and 2.00 mg/cm2 (± 10%) per the randomization schedule using a 1cc tuberculin syringe (without a needle) or pipette and a clean finger cot for approximately 20 to 50 seconds.
  Interventions: Other: Sunscreen A
- Sunscreen B (Experimental): At each visit, each enrolled subject will be randomly assigned 1 of the 3 Sunscreens to apply to both lower legs (between the knee and ankle) and then her full face. The subject will cleanse her hands with soap and water between the lower legs and face Sunscreen applications.
  After lower legs and facial Sunscreen applications are completed, a trained designee will delineate six 4 cm x 4 cm test sites on the subject's volar forearms (3 test sites per volar forearm). Then a trained designee will apply the assigned Sunscreen to the designated test sites in a consistent manner at a randomly assigned dose density of 0.25, 0.50, 0.75, 1.00, 1.50, and 2.00 mg/cm2 (± 10%) per the randomization schedule using a 1cc tuberculin syringe (without a needle) or pipette and a clean finger cot for approximately 20 to 50 seconds.
  Interventions: Other: Sunscreen B
- Sunscreen C (Experimental): At each visit, each enrolled subject will be randomly assigned 1 of the 3 Sunscreens to apply to both lower legs (between the knee and ankle) and then her full face. The subject will cleanse her hands with soap and water between the lower legs and face Sunscreen applications.
  After lower legs and facial Sunscreen applications are completed, a trained designee will delineate six 4 cm x 4 cm test sites on the subject's volar forearms (3 test sites per volar forearm). Then a trained designee will apply the assigned Sunscreen to the designated test sites in a consistent manner at a randomly assigned dose density of 0.25, 0.50, 0.75, 1.00, 1.50, and 2.00 mg/cm2 (± 10%) per the randomization schedule using a 1cc tuberculin syringe (without a needle) or pipette and a clean finger cot for approximately 20 to 50 seconds.
  Interventions: Other: Sunscreen C

INTERVENTIONS:
Other: Sunscreen A — Sunscreen A will be applied to both lower legs (between the knee and ankle) and then her full face to the randomly assigned participants at Visit1, Visit 2, and Visit 3.
  Arms: Sunscreen A
Other: Sunscreen B — Sunscreen B will be applied to both lower legs (between the knee and ankle) and then her full face to the randomly assigned participants at Visit1, Visit 2, and Visit 3.
  Arms: Sunscreen B
Other: Sunscreen C — Sunscreen C will be applied to both lower legs (between the knee and ankle) and then her full face to the randomly assigned participants at Visit1, Visit 2, and Visit 3.
  Arms: Sunscreen C

SUMMARY:
The purpose of the study is to evaluate the whitening potential of different mineral and chemical sunscreens across multi-cultural skin tones through instrumentation, imaging, and self-assessment. It also aimed to evaluate the relationship between self-perception and objective measurements of whitening.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported natural skin tone/skin color targeting the following: skin tones "Pale/fair to light white" and "White to light beige" (N = 15 participants), skin tones "Beige to light tan/light olive" and "Medium tan/medium olive to light brown" (N = 15 participants), skin tones "Medium brown to dark brown and "Darkest brown to darkest black" (N = 15 participants)
* Has a history of using or is a current user of sunscreens
* Is willing to have height and body weight measured and recorded
* Generally in good health based on medical history reported by the participants
* Is able to read, write, speak, and understand English or Spanish
* Has signed the ICD including Health Insurance Portability and Accountability Act (HIPAA) disclosure and Photograph Release
* Intends to complete the study and is willing and able to follow all study instructions

Exclusion Criteria:

* Has known allergies or adverse reactions to common topical skincare products or ingredients in the IPs
* Presents with a skin condition and/or pre-existing or dormant dermatologic disease on the face, volar forearms, or lower legs that may confound the study results (e.g., psoriasis, eczema, atopic dermatitis, cutaneous xerosis, erythema, or active skin cancer, rosacea, moderate to severe acne, acne conglobate, nodules, and/or cysts on the face) or interfere with evaluations (e.g., excessive hair, tattoos, scarring, nevi, very uneven skin tone, sunburn, scratches/broken/compromised skin)
* Has had any facial treatments including facials, facial peels, photo facials, laser treatments, dermabrasion, botulinum toxin (Botox), injectable filler treatments, intense pulsed light (IPL), acid treatments, tightening treatments, facial plastic surgery, or any other treatment administered by a physician or skin care professional designed to improve the appearance or firmness of facial skin withing 30 days prior to Visit 1
* Has shaved or used any hair removal method on lower legs or volar forearms within 24 hours of Visit 1
* Has a history of skin cancer within the past 5 years
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication
* Is taking a medication that would mask an Adverse Event (AE) or confuse the study results
* Has a history of immunosuppression/immune deficiency disorders (including HIV infection, AIDS, multiple sclerosis, Crohn's disease, rheumatoid arthritis), organ transplant (heart, kidney, etc.), and/or undergoing radiation or chemotherapy as determined by study documentation
* Has a disease such as asthma, epilepsy, hypertension, hyperthyroidism, or hypothyroidism that is not controlled by diet or medication. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc.
* Is self-reported to be breast feeding, pregnant or planning to become pregnant during the study
* Has a history of or a concurrent health/other condition/situation which may put the individual at significant risk, confuse the study results, or interfere significantly with the individual's participation in the study
* Has started any long-term medication within the last 2 months
* Is simultaneously participating in any other clinical study or has participated in any product-use study within 30 days prior to Visit 1
* Is an employee/contractor or immediate family member of the PI, Study Site, or Sponsor

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Whitening Potential of Mineral Sunscreens Across Multi-cultural Skin Tones Through Instrumentation | Visit 1 (Day 1), Visit 2 (Day 7) and Visit 3 (Day 14)
  Whitening potential of mineral sunscreens across multi-cultural skin tones through instrumentation (Chroma Meter and Polychromatic Hybrid Diffuse Reflectance Spectroscopy measurements) will be reported.
Whitening Potential of Mineral Sunscreens Across Multi-cultural Skin Tones Through Imaging | Visit 1 (Day1), Visit 2 (Day 7) and Visit 3 (Day 14)
  Whitening potential of mineral sunscreens across multi-cultural skin tones through imaging (Full-Face Imaging via VISIA-CR and Volar Forearms Imaging via Digital Camera) will be reported.
Whitening Potential of Mineral Sunscreens Across Multi-cultural Skin Tones Through Self-assessment | Visit 1 (Day1), Visit 2 (Day 7) and Visit 3 (Day 14)
  Whitening potential of mineral sunscreens across multi-cultural skin tones through self-assessment will be reported via self-assessment questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- SGS North America Inc. - Union Research Center, Union, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No